CLINICAL TRIAL: NCT03139617
Title: Comparison the Efficacy as Analgesia Between Ultrasound Guided Femoral 3 in 1 Block Versus Blind Fascia Iliaca Block for Positioning Prior Spinal Anaesthesia in Femur Fracture Surgery
Brief Title: Comparison Between Ultrasound Guided Femoral 3 in 1 Block Versus Blind Fascia Iliaca Block Before Spinal Anaesthesia
Acronym: IKH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rhendra Hardy Mohamad Zaini, Doctor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/15100313
Record Dates: First submitted 2017-04-15; First posted 2017-05-04 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Regional Anaesthesia
Keywords: Fascia Iliaca Block; Femoral 3-in-1 block; Fracture femur; Spinal anesthesia
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fascia Iliaca Compartment Block (FICB) (Active Comparator): fascia iliaca compartment block is done using a blind technique with a blunt size 24 Gauge (G) needle. The technique is based upon the anatomical landmark and once located the space local anaesthetic ropivacaine 0.375% will be given based on the body weight.
  Interventions: Procedure: Fascia Iliaca Compartment Block (FICB)
- 3 in 1 femoral block (FNB) (Experimental): Ultrasound guided femoral 3 in 1 block using insulated stimulating needle 22 Gauge (G). Ropivacaine 0.375% as per ideal body weight.
  Interventions: Procedure: 3 in 1 femoral block (FNB)

INTERVENTIONS:
Procedure: Fascia Iliaca Compartment Block (FICB) — The FICB was done in the OT with standard monitoring with emergency airway intervention and resuscitation drug prepared before performing intended block. Patient was put in supine position, using aseptic technique, chlorhexidine solution and draped with sterile medical towel. Lignocaine 2% for local anaesthetic infiltration at punctured site.A blunted needle (Plexufix® 24G x 2", B Braun Melsungen AG 34209 Germany).A line was drawn from pubic tubercle to anterior superior iliac spine, the punctured point is 2-3cm distal to the point where medial 2/3rd and lateral 1/3rd of the line meet. Loss of resistance 2 times indicated the punctured of fascia lata and iliaca.A total volume of Ropivacaine 0.375% per body weight was given with repeated aspiration.
  Arms: Fascia Iliaca Compartment Block (FICB)
Procedure: 3 in 1 femoral block (FNB) — The FNB was done in the OT with standard monitoring with emergency airway intervention and resuscitation drug prepared before performing intended block.Patient was put in supine position, using aseptic technique, chlorhexidine solution and draped with sterile medical towel.Lignocaine 2% for local anaesthetic infiltration at punctured site.An insulated stimulating needle (Stimuplex® D Plus 22g x 2", B Braun Melsungen AG 34209 Melsungen Germany). Ultrasound was used to locate the femoral vessel and nerve and by using 'in plane' technique, the skin was punctured with the insulated needle and advance in transverse plane at around 30 angle to the skin. Local anaesthetic solution as per ideal body weight given after negative aspiration of blood .
  Arms: 3 in 1 femoral block (FNB)

SUMMARY:
This study aimed to evaluate the efficacy of ultrasound guided femoral 3 in 1 block versus the blind technique single shot fascia iliaca compartment block as an analgesia method in patients prior positioning for spinal anaesthesia in femur fracture surgery. A total of 60 patients were enrolled and divided equally into 2 groups.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy of fascia iliaca compartment block comparing to femoral nerve block. If it is proven effective, this technique should be implemented as a method of analgesia (pain relief) prior positioning for spinal anaesthesia. As fascia iliaca compartment block is relatively easy to be done without the need of advanced equipment, it has the potential role for good pain management in patient with femur fracture. Thus this will reduce the need of intravenous or oral analgesic such as opioid or nonsteroidal anti-inflammatory drugs and side effects that comes with it.

This is a prospective single blind randomized study of a total of 60 patients ASA I - III who were scheduled to undergo fixation of femur fractures. Patients who fulfilled the criteria were recruited after informed consent was taken. This study was conducted in the operation theatres of the Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan.

Hypothesis

1. There is no difference in term of success rate between ultrasound guided Femoral 3 in 1 nerve block versus Single shot blind Fascia Iliaca Compartment Block prior positioning for spinal anaesthesia in femur fracture surgery.
2. There is no difference in term of analgesic effect between ultrasound guided Femoral 3 in 1 nerve block versus Single shot blind Fascia Iliaca Compartment Block prior positioning for spinal anaesthesia in femur fracture surgery.
3. There is no different in term of onset of analgesia between Femoral 3 in 1 nerve block versus Fascia Iliaca Compartment Block prior positioning for spinal anaesthesia in femur fracture surgery.

Recruitment and Randomization Eligible patients will be approach and offered to participate in this study prior operation. Agreed patients will have to sign informed consent Subject will be randomized into 2 groups using computer assisted randomization

Sample Size Calculation The sample size was calculated based on reduction of visual analog score in a study done by Newman et al with score 3.7±2.6, α = 0.05 and power of study 80%. The patients were randomized per a computerized generated random number and divided into two groups. Group A (FICB) n = 30, received single shot fascia iliaca compartment block (blind technique) and the other group B (FNB) n = 30 received ultrasound guided femoral 3 in 1 block. Initial target sample of 66 was calculated including drop out, however as there was no drop out from the study we decided to stop at 60 samples only. As 30 samples for each arm was adequate for a clinical study to be conducted and data acquired can be statistically analysed.

Study Protocol After ethic approval, written informed consent will be obtained from participants that met inclusion/exclusion criteria.

A total of 66 adults who are planned for open reduction internal fixation (ORIF) of proximal femur fracture will be enrolled. Easy sample random sampling using opaque and sealed envelope will be used to divide patient into Group 1 (Group Femoral 3 in 1 Block) and Group 2 (Fascia Iliaca Compartment Block) with ratio 1:1.

Random sampling will be done upon patient arrival to reception area in operation theatre complex. Both block will be performed by principal investigator in induction anaesthetic room while waiting for surgery. Data will be collected by registered nurse anaesthetist monitoring preoperatively and resident anaesthetist who's in charge in the operating theatre.

Block will be performed in induction room near the recovery area in operating theatre (OT) complex. Basic and standardized monitoring as listed by American Society of Anaesthesiologist (ASA) will be applied such as Non-invasive blood pressure monitoring (NIBP), Heart rate (HR), Oxygen saturation (SpO2) and electrocardiogram (ECG). Patient will be monitored continuously during the procedure. Apart from that, a variable performance oxygen delivery system will be given using nasal cannula at 3 litre/min. At least 1 functioning cannula will be made available with running IV drip. Preparation for emergency airway intervention and resuscitation drug will also be prepared before performing intended block.

In both group, block will be performed with patient in supine position, under aseptic technique using chlorhexidine solution and drape with sterile medical towel. Both group will be given Lignocaine 2% for local infiltration at puncture site. Ropivacaine 0.375% will be used in both groups with a total volume depends on weight basis.

Group 1 (Femoral 3 in 1 Block/FNB) This group will be given femoral 3 in 1 block Needle: Stimuplex or Locoplex 22-gauge 50-mm insulated needle Using Ultrasound guidance and peripheral nerve stimulator. Total Volume of Local anaesthetic: 20-40mls. Ultrasound will be use to locate the femoral vessel and nerve. Using 'in plane' technique, the needle will be puncture and advance in transverse plane at a 30 angle to the skin. Peripheral Nerve stimulator will be used if there is difficulty in recognizing the nerve, stimulation of the nerve will cause contraction of quadriceps femoris muscle. A total 20-40mls of local anaesthetic solution as per ideal body weight will be injected over a 2-3minutes duration after careful negative aspiration of blood to rule out inadvertent intravascular puncture. Careful aspiration will be done in every 3-5mls injection until a total of 20-40mls local anaesthetic being delivered.

Group 2: Fascia Iliaca Compartment Block (FICB) This group will be given fascia iliaca compartment block as shown in figure 3. Needle: Luer Lock cannula (Plexufix) 24-gauge 50-mm insulated needle Total Volume of Local anaesthetic: 20-40mls based on ideal body weight The technique is done as described by Dalens et al, 1989 using anatomical landmark technique. A line is drawn from pubic tubercle to anterior superior iliac spine (ASIS) and divided into 3 equal parts. The puncture point is 2-3cm distal to the point where medial 2/3rd and lateral 1/3rd of the line meet. The femoral vessel will be identified and should lie medial to the puncture site. The fascia iliaca block will be perform without using the nerve stimulator or ultrasound.

By using a blunted needle (24G, plexufix needle), identification of puncturing intended space is by feeling 2 times loss of resistance (described as clicks or plops). This indicates the puncture of fascia lata and fascia iliaca. After careful aspiration with syringe to rule out inadvertent vascular injection, a total volume of local anaesthetic (LA) will be given according to group allocation and body weight. Bolus of LA given in 2-3minutes duration with repeated aspiration. In case of accidental vascular puncture, needle is withdrawn and punctured site will be compressed for 5 minutes to avoid haematoma before reattempt lateral 1-2cm from initial site.

For both group, any signs of complication will be look for, documented and treated accordingly. Examples are:

1. Local anaesthetic toxicity such tingling sensation around mouth, metallic taste, light headache, confusion, altered conscious level, seizures, visual disturbances, arrhythmias and cardiovascular collapse
2. Swelling at site of puncture due to hematoma or localization of local anaesthetic
3. Bleeding from puncture site

Precaution to avoid complication from procedure:

1. Dose local anaesthetic should be precalculated to avoid toxicity, total maximum dose of Ropivacaine is 3mg/kg
2. Careful negative aspiration before giving intended local anaesthetic in titrating dose to avoid inadvertent vascular puncture
3. Total volume of local anaesthetic given in repeated aspiration and in titrating dose in 2-3 minutes' duration

ELIGIBILITY:
Inclusion Criteria:

* ASA I - III with stable hemodynamic parameters
* Planned for open reduction internal fixation of fracture femur under spinal anaesthesia

Exclusion Criteria:

* Coagulopathy/ Bleeding diathesis
* Known allergy to amide local anaesthetic used in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The percentage of success rate between ultrasound guided femoral 3 in 1 block versus single shot blind fascia iliaca compartment block as analgesic method for positioning prior spinal anaesthesia in femur fracture surgery | From the time of local anaesthetic injection to successful block at least 2 out of 3 dermatomes of either lateral femoral cutaneous nerve, femoral nerve or obturator nerve up to 30 minutes.
  Using pin prick to test the sensory level at different dermatomes after given local anaesthetic following each block

SECONDARY OUTCOMES:
The onset of analgesia in term of minutes between ultrasound guided Femoral 3 in 1 nerve block versus single shot blind Fascia Iliaca Compartment Block prior positioning for spinal anaesthesia in femur fracture surgery. | From the time of local anaesthetic given to a reduction in visual analogue pain score to less than 2 up to 30 minutes.
  assessment of the patient pain severity post local anaesthetic injection after each block by using the visual analogue pain score chart
The quality of blocks | From the sitting up the patients till successful spinal anesthesia was achieved up to 10 minutes.
  The quality of positioning the patients documented by the operator prior to giving spinal anaesthesia level

CONTACTS AND LOCATIONS:
Overall Officials: Rhendra Hardy Mohamad Zaini, MD, Principal Investigator — Universiti of Science Malaysia
Locations (1):
- University of Science Malaysia Hospital, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lopez S, Gros T, Bernard N, Plasse C, Capdevila X. Fascia iliaca compartment block for femoral bone fractures in prehospital care. Reg Anesth Pain Med. 2003 May-Jun;28(3):203-7. doi: 10.1053/rapm.2003.50134. PMID 12772137
- [Result] Capdevila X, Biboulet P, Bouregba M, Barthelet Y, Rubenovitch J, d'Athis F. Comparison of the three-in-one and fascia iliaca compartment blocks in adults: clinical and radiographic analysis. Anesth Analg. 1998 May;86(5):1039-44. doi: 10.1097/00000539-199805000-00025. PMID 9585293
- [Result] Winnie AP, Ramamurthy S, Durrani Z. The inguinal paravascular technic of lumbar plexus anesthesia: the "3-in-1 block". Anesth Analg. 1973 Nov-Dec;52(6):989-96. No abstract available. PMID 4796576
- [Result] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650